CLINICAL TRIAL: NCT00665821
Title: Study of the Effect of Two Short Education Programs for the Treatment of Nonspecific Low Back Pain in Patients Seen at a Workers' Health Care Organization
Brief Title: The Effect of Two Short Education Programs for Nonspecific Low Back Pain in a Workers' Health Care Organization
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: From Sept./08 to April/09 only 30 subjects were recruited. It has proved extremely difficult to recruit subjects.
Sponsor: Kovacs Foundation (Other)
Collaborators: Hospital Laboral SOLIMAT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FK-S-24
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain
Keywords: nonspecific low back pain; disability; sick leave; catastrophizing; workers
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Classic back pain prevention education, and cognitive behavioral management. — Classic education: postural hygiene, Back Guide. Cognitive behavioral management: active management, Back Book.
Behavioral: General health education — General health education: a booklet describing general norms for maintaining good health

SUMMARY:
The purpose of this study is to assess the effect of two different types of health education programs on the disability, beliefs related to low back pain and duration of sick leave in patients seen at a workers' health care organization

ELIGIBILITY:
Inclusion Criteria:

* low back pain patients, with or without referred or radiated pain
* no systemic disease or criteria for referral to surgery

Exclusion Criteria:

* inability to fill out the questionnaires and scales
* bedridden
* rheumatologic inflammatory disease, cancer or fibromyalgia
* suspicion of fibromyalgia
* spinal fracture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2008-09; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
A reduction in low back pain related disability and sick leave. | 365 days

SECONDARY OUTCOMES:
A reduction in catastrophizing beliefs related to low back pain. | 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Andrés Barriga, MD, Principal Investigator — Hospital Laboral Solimat, Toledo, Spain
Locations (2):
- Spain (2):
  - Kovacs Foundation, Palma de Mallorca, Balearic Islands
  - Hospital Laboral SOLIMAT, Toledo, Castille-La Mancha

REFERENCES:
- [Background] Burton AK, Waddell G, Tillotson KM, Summerton N. Information and advice to patients with back pain can have a positive effect. A randomized controlled trial of a novel educational booklet in primary care. Spine (Phila Pa 1976). 1999 Dec 1;24(23):2484-91. doi: 10.1097/00007632-199912010-00010. PMID 10626311
- [Background] Frost H, Lamb SE, Doll HA, Carver PT, Stewart-Brown S. Randomised controlled trial of physiotherapy compared with advice for low back pain. BMJ. 2004 Sep 25;329(7468):708. doi: 10.1136/bmj.38216.868808.7C. Epub 2004 Sep 17. PMID 15377573
- [Background] Kovacs F, Abraira V, Santos S, Diaz E, Gestoso M, Muriel A, Gil del Real MT, Mufraggi N, Noguera J, Zamora J; Spanish Back Pain Research Network. A comparison of two short education programs for improving low back pain-related disability in the elderly: a cluster randomized controlled trial. Spine (Phila Pa 1976). 2007 May 1;32(10):1053-9. doi: 10.1097/01.brs.0000261556.84266.0f. PMID 17471084